CLINICAL TRIAL: NCT00869141
Title: Earlier Intraocular Pressure Control After Ahmed Glaucoma Valve Implantation for Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Simon Law, Clinical Associate Professor of Health Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCLA IRB#08-10-110-01
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-07

CONDITIONS: Glaucoma
Keywords: Glaucoma tube shunt procedure
MeSH Terms: conditions — Glaucoma | interventions — Timolol; Brimonidine Tartrate; dorzolamide; brinzolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Research arm (postop IOP>10) (Experimental): Receive glaucoma medications if the eye pressure more than 10 mmHg after AHmed valve implantation
  Interventions: Drug: glaucoma medications (Timolol, Brimonidine, Dorzolamide, Brinzolamide)
- Standard of care arm (postop IOP>17) (Active Comparator): Receive glaucoma medication if eye pressure more than 17 mmHg after Ahmed valve implantation
  Interventions: Drug: glaucoma medications (Timolol, Brimonidine, Dorzolamide, Brinzolamide)

INTERVENTIONS:
Drug: glaucoma medications (Timolol, Brimonidine, Dorzolamide, Brinzolamide) — Subjects may receive glaucoma medications after Ahmed valve implantation
  Other Names: Timolol, Brimonidine, Dorzolamide, Brinzolamide

SUMMARY:
The purpose of this study is to compare the occurrence rate of the high pressure phase and the final pressure outcomes between patients treated with glaucoma medication prior to the expected onset of the high pressure phase to those patients who have glaucoma medication started at the onset of the high pressure phase. The investigators hypothesize that if glaucoma medications are started prior to the expected onset of high pressure phase, the high pressure phase will not occur as frequently and the ultimate pressure level will be lower than if the glaucoma medications are started at the onset of this phase.

DETAILED DESCRIPTION:
Tube shunt procedures are a popular surgery for the control of glaucoma. Tube shunt devices are designed to drain eye fluid (aqueous humor) through a tube inserted into the front chamber of the eye (anterior chamber) to a plate secured to the mid-posterior section of the outer eyeball wall. The body then lays down collagen tissue and forms a capsule around the plate. The fluid filters through the capsule of collagen tissue and is reabsorbed into the ocular and systemic circulation. The collagen tissue continues to remodel itself over a long period of time (up to years). However, a well characterized, yet poorly understood, phenomenon occurs in many patients in the 4-8 weeks after the device's implantation, called the hypertensive phase. The pressure of the eye can increase from a desirable level of about 10 immediately after the tube shunt implantation to much higher levels, in the range of 20 to 30's, and then it may gradually return to less than 20. Such a high pressure phase can cause irreversible damage an eye with glaucoma. The usual management of a high pressure phase is to start glaucoma medications as soon as it is detected. A previous study we conducted showed that this high pressure phase resolves in about half of patients with medical therapy, but the other half may continue to have higher than expected pressures. The exact cause of this high pressure phase is unknown. However, it is postulated that the mechanism may involve a compaction collagen tissue layers under the eye's own fluid pressure while the collagen tissue is being laid down, which in turn creates a firm, dense capsule that makes escape of fluid difficult. Therefore, it is argued that if the formation of eye fluid is reduced by medication during this initial period when the collagen tissue is laid down, the compaction of collagen, and subsequently the high pressure phase may be avoided.

The purpose of this study is to compare the occurrence rate of the high pressure phase and the final pressure outcomes between patients treated with glaucoma medication prior to the expected onset of the high pressure phase to those patients who have glaucoma medication started at the onset of the high pressure phase. We hypothesize that if glaucoma medications are started prior to the expected onset of high pressure phase, the high pressure phase will not occur as frequently and the ultimate pressure level will be lower than if the glaucoma medications are started at the onset of this phase.

We believe that this study will have a very significant impact on the management of glaucoma with tube shut procedures. If it is true that the rate and pressure level of the hypertensive phase can be reduced by simply starting glaucoma medications to reduce the formation of eye fluid before the expected the high pressure phase begins, which is generally 4 weeks after implantation of the tube shunt device, glaucoma patients can be saved from exposure to the very high level of eye pressure, and the eventual pressure control may be better.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring Ahmed glaucoma valve implantation to control intraocular pressure between the ages of 18 and 85 years.

Exclusion Criteria:

1. Unwilling or unable to give consent or unwilling to accept randomization.
2. Patient out of area and potentially unavailable for follow-up visits.
3. Known allergic reaction to timolol, brimonidine, dorzolamide, brinzolamide, or sulfa drugs.
4. Known medical contraindications to the use of beta-blockers, including congestive heart failure, heart block, asthma, and chronic obstructive pulmonary disease.
5. Concurrent intraocular procedure with Ahmed glaucoma valve implantation
6. Previous Ahmed glaucoma valve implantation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon K Law, MD, Principal Investigator — Jules Stein Eye Institute, University of California Los Angeles
Locations (1):
- Juels Stein Eye Institute, Los Angeles, California, United States

REFERENCES:
- See also: Jules Stein Eye Institute — http://www.jsei.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Research Arm: Receive glaucoma medications if the eye pressure more than 10 mmHg after AHmed valve implantation
  glaucoma medications (Timolol, Brimonidine, Dorzolamide, Brinzolamide): Subjects may receive glaucoma medications after Ahmed valve implantation
- Standard of Care Arm: Receive glaucoma medication if eye pressure more than 17 mmHg after Ahmed valve implantation
  glaucoma medications (Timolol, Brimonidine, Dorzolamide, Brinzolamide): Subjects may receive glaucoma medications after Ahmed valve implantation
Period: Overall Study
Arm/Group | Research Arm | Standard of Care Arm
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Research Arm | Standard of Care Arm | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (11.6) | 61.6 (15.3) | 64.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 13 | 15 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 23 | 21 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 10 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Hypertensive Phase After Ahmed Valve Implantation for Glaucoma
Description: Intraocular pressure more than 21 mmHg during the first 6 months after Ahmed valve implantation after the pressure has been reduced to less than 22 mmHg in the first postoperative week
Time Frame: within 6 months after surgery
Measure: Number; unit: participants
Arm/Group | Research Arm | Standard of Care Arm
Number analyzed (Participants) | 26 | 26
participants | 9 | 12

2. Primary Outcome: Intraocular Pressure Control After Ahmed Valve Implantation for Glaucoma
Description: intraocular pressure comparison between groups after the Ahmed valve implantation
Time Frame: 3 weeks after surgery
Population: Eye pressure at postop 3-week is reported
Measure: Mean (Standard Deviation); unit: mmHg at postop 3-week
Arm/Group | Research Arm | Standard of Care Arm
Number analyzed (Participants) | 26 | 26
mmHg at postop 3-week | 15.6 (3.6) | 20.6 (8.9)

3. Primary Outcome: Intraocular Pressure of Eyes With Hypertensive Phase Versus Without Hypertensive Phase
Description: intraocular pressure of eyes with hypertensive phase versus without hypertensive phase
Time Frame: 1 year after surgery
Population: Please note that these two groups were different from those groups in previous comparison. The patients that developed hypertensive phase were compared to those that did not developed hypertensive phase, so the number of patients in these two groups and the mean pressure at 1 year +/-standard deviation results were different.
Measure: Mean (Standard Deviation); unit: mmHg in 1 year postop
Groups:
- Hypertensive Phase Group: Eyes that developed hypertensive phase after Ahmed valve implantation
- Non-hypertensive Phase Group: Eyes that did not develop hypertensive phase after Ahmed valve implantation
Arm/Group | Hypertensive Phase Group | Non-hypertensive Phase Group
Number analyzed (Participants) | 21 | 31
mmHg in 1 year postop | 15.1 (5.2) | 11.4 (4.3)

ADVERSE EVENTS:
Arm/Group | Research Arm | Standard of Care Arm
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 1/26 | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Research Arm (N=26) | Standard of Care Arm (N=26)
Uveitis and conreal edema (Eye disorders) | 0 (0) | 2 (2)
Strabismus (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No